CLINICAL TRIAL: NCT04530084
Title: A Single Center Proof Of Concept Study To Assess Intra And Perioperative Safety Profile Of OMNI Surgical System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mark Gallardo, MD (Other)
Responsible Party: Sponsor-Investigator, Mark Gallardo, MD, Principal Investigator, El Paso Eye Surgeons
Organization: El Paso Eye Surgeons (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1290569
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Diagnosed with open angle glaucoma (Experimental)
  Interventions: Device: OMNI Surgical System

INTERVENTIONS:
Device: OMNI Surgical System — Scheduled for canaloplasty and trabeculotomy with or without cataract extraction

SUMMARY:
The overall objective of this study is to determine the safety and usability of OMNI surgical system in performing canaloplasty and trabeculotomy. Outcome measures will include 1) adverse events (intraoperative and perioperative) 2) BCVA 3) Secondary surgical interventions 4) mean IOP and 5) mean number of hypotensive medications

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 22 years or older.
2. Visually significant cataract or pseudophakic with a posterior chamber intraocular lens (PCIOL)
3. Diagnosed with open angle glaucoma (e.g. primary open angle glaucoma, pigmentary glaucoma, pseudoexfoliative glaucoma)
4. Scheduled for canaloplasty and trabeculotomy

Exclusion Criteria:

1. Any other intraocular surgery at the time of canaloplasty and trabeculotomy excepting cataract surgery for those subjects with cataract.
2. Prior trabeculectomy, other bleb-forming glaucoma surgery (e.g. tube shunt), or implanted trabecular bypass stents.
3. Any other ocular pathologies that may interfere with the study procedure or be exacerbated by the OMNI procedure.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-08-21 (Actual); Primary Completion 2021-08-22 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events (intraoperative and perioperative) | 3 months
Best Corrected Visual Acuity (BCVA) | 3 months

SECONDARY OUTCOMES:
Mean intraocular pressure (IOP) | 3 months
Mean number of ocular hypotensive medications | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- El Paso Eye Surgeons, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No